CLINICAL TRIAL: NCT03823924
Title: Body Composition and Bone Mineral Density in Patients With Psoriatic Arthritis and Changes After 6 Months of Treatment With Ustekinumab
Brief Title: Changes in Body Composition Under Ustekinumab in PsA
Acronym: STELARA-CC
Status: Terminated | Type: Observational
Why Stopped: logistic problems
Sponsor: University Hospital, Lille (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017_39; 2018-A01552-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-14; First posted 2019-01-31 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2021-09

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; ustekinumab; body composition; bone mineral density; adiposity
MeSH Terms: conditions — Arthritis, Psoriatic; Obesity | interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psoriatic arthritis
  Interventions: Procedure: Bone mineral density (BMD)
- Healthy volunteers
  Interventions: Procedure: Bone mineral density (BMD)

INTERVENTIONS:
Procedure: Bone mineral density (BMD) — The bone mineral density (BMD) performed by DXA, which will allow the analysis of bone density (mg / cm²) at the lumbar spine (BMD L1 to L4) and the total hip (non-dominant).
  This examination will also allow an analysis of the body composition at the same time (lean mass, fat mass and bone mass for the whole body).

SUMMARY:
There is not much body composition and bone mineral density data available for patients with psoriatic arthritis (rheumatoid arthritis) compared to control subjects.

The evaluation of the total fat mass and in particular of its abdominal distribution (visceral adiposity) is important because an excessive adiposity generates adverse effects on the health (hypertension, dyslipidemia, cardiovascular risk and resistance to the insulin).

In addition, data on changes in body composition and bone mineral density were not available under a new psA treatment, namely ustekinumab (anti-IL12 / 23 antibody).

It is proposed to conduct a pilot study to evaluate body composition, distribution (visceral adiposity) and bone mineral density in patients with psoriatic arthritis (versus control subjects) and their changes after 6 months of treatment with ustekinumab

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic arthritis:

  1. Men and women ≥ 18 years
  2. Patients with PsA according to CASPAR criteria,
  3. Patients who do not have yet started ustekinumab,
  4. Patients who signed the informed consent.
* Healthy volunteers:

  1. Men and women ≥ 18 years
  2. Patients who signed the informed consent.

     Exclusion Criteria:
* Items 1 to 10 are applicable to healthy volunteers and PsA

  1. History of fragility fracture AND / OR T-score ≤-3 if ≥50 years AND / OR Z-score ≤-3 if <50 years during the screening phase,
  2. Corticosteroids ≥10 mg / day,
  3. Diseases or treatments affecting bone metabolism (breast cancer with anti-aromatase, malabsorption, primary hyperparathyroidism, uncontrolled hyperthyroidism ...),
  4. History of radiotherapy on the lumbar spine or hip,
  5. Patients undergoing hormone replacement therapy (HRT) or patients already on anti-osteoporotic therapy (bisphosphonates, strontium ranelate, teriparatide or denosumab),
  6. Chronic kidney disease with creatinine clearance (CKD-EPI) ≤ 30 ml / min,
  7. Weight> 160 kg,
  8. Patients under restrictive diet or considering a diet of this type during the study period,
  9. Patients who have an intense exercise program or plan to benefit from it during the study period,
  10. Pregnant or lactating women or having a pregnancy project,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with psoriatic arthritis and controls
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-07-11 (Actual)

PRIMARY OUTCOMES:
Visceral adiposity (VAT) | At baseline
  Comparison at baseline of visceral adiposity (VAT) in cm² between PsA (n = 30) and healthy volunteers (n = 30) matched on age (± 5 years, ≥ 18 years), sex, menopausal status for women and body mass index (BMI, ± 3 kg / m²).

SECONDARY OUTCOMES:
Total lean mass | At baseline
  Comparison at baseline of total lean mass (TLM, kg), between PsA (n = 30) and healthy volunteers (n = 30) matched on age (± 5 years, ≥ 18 years), sex, menopausal status for women and body mass index (BMI, ± 3 kg / m²).
Total fat mass | At baseline
  Comparison at baseline of total fat mass (TBF, %) between PsA (n = 30) and healthy volunteers (n = 30) matched on age (± 5 years, ≥ 18 years), sex, menopausal status for women and body mass index (BMI, ± 3 kg / m²).
Bone mineral density | At baseline
  Comparison at baseline of bone mineral density (BMD, g/cm²) between PsA (n = 30) and healthy volunteers (n = 30) matched on age (± 5 years, ≥ 18 years), sex, menopausal status for women and body mass index (BMI, ± 3 kg / m²).
Change in total fat mass (TBF, %) under ustekinumab in PsA | at baseline and at 6 months (± 2 months)
Change in total lean mass (TLM, kg) under ustekinumab in PsA | at baseline and at 6 months (± 2 months)
Change in visceral adiposity (cm²) under ustekinumab in PsA | at baseline and at 6 months (± 2 months)
Change in bone mineral density (BMD, g/cm²) under ustekinumab in PsA | at baseline and at 6 months (± 2 months)
Change in makers of bone remodeling under ustekinumab in PsA | at baseline and at 6 months (± 2 months)
  C-telopeptide (Ctx), Procollagen type 1 amino-terminal propeptide (P1NP)
Change in leptin under ustekinumab in PsA | at baseline and at 6 months (± 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Julien Paccou, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France